CLINICAL TRIAL: NCT00517582
Title: Study of a Bradykinin Receptor Blocker in Angiotensin Converting Enzyme Inhibitor-Associated Angioedema
Brief Title: Bradykinin Receptor Blocker in ACE Inhibitor-associated Angioedema
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was stopped to allow initiation of a mult-center study
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 495; R01HL079184 (NIH); HL079184-Specific Aim 1
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Angioneurotic Edema
Keywords: ACE Inhibitor; Angioedema; Bradykinin; Swelling
MeSH Terms: conditions — Angioedema | interventions — icatibant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOE-140 (Experimental): Administration of HOE-140 (icatibant) 30 mg at time 0 and at 6 hours
  Interventions: Drug: HOE-140
- Placebo (Placebo Comparator): Administration of placebo at time 0 and 6 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HOE-140 — Subcutaneous at time 0 and 6 hours
  Other Names: icatibant
  Arms: HOE-140
Other: Placebo — Subcutaneous at time 0 and 6 hours
  Arms: Placebo

SUMMARY:
Individuals with heart disease or high blood pressure are often prescribed angiotensin converting enzyme (ACE) inhibitors to treat their disease. However, the use of ACE inhibitors can be associated with angioedema, a rare but life-threatening condition that causes swelling of the face and other body parts. This study will evaluate the effectiveness of the drug HOE-140 at decreasing symptoms of angioedema in people taking ACE inhibitors who develop the condition.

DETAILED DESCRIPTION:
People who take ACE inhibitors may develop angioedema, a condition that causes itchy and painful swelling beneath the skin around the eyes, lips, tongue, throat, hands, or feet. In severe cases, the throat may swell, obstructing the airway and leading to breathing difficulty. ACE inhibitors prevent the breakdown of a natural chemical in the body called bradykinin. Increased levels of bradykinin, which can cause swelling, may contribute to the development of angioedema. Blocking bradykinin receptor cells prevents bradykinin from initiating swelling and may lead to a possible decrease in angioedema symptoms. The purpose of this study is to evaluate the effectiveness of HOE-140, a bradykinin receptor blocker, at reducing symptoms in people with ACE inhibitor-associated angioedema.

This study will enroll people admitted to the emergency room or hospital who have a severe case of ACE inhibitor-associated angioedema. Participants will be randomly assigned to receive an injection of either HOE-140 or placebo. Initially, participants will undergo an electrocardiogram to measure the electrical activity of the heart. Then blood pressure measurements, blood collection, a physical exam to determine the extent and duration of swelling, and photographs of the swelling will occur at 2, 4, 8, 16, and 24 hours following the start of treatment. Questionnaires will be completed by study staff and participants to assess changes in angioedema symptoms and the extent of swelling. Participants will remain in the hospital for 24 to 48 hours, depending on the severity of their symptoms. Blood will be collected at a follow-up visit that will occur 7 days after the resolution of angioedema symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* ACE inhibitor-associated angioedema, as defined as swelling of the lips, pharynx, or face while taking an ACE inhibitor, no history of angioedema while not taking an ACE inhibitor, and no evidence of abnormal C1 inhibitor concentration or abnormal complement levels. People with possible cases of ACE inhibitor-associated bowel edema will not be enrolled.
* If female, must be postmenopausal for at least 1 year prior to study entry, undergone surgical sterilization, or willing to use an effective form of birth control and take a pregnancy test daily for the duration of the study

Exclusion Criteria:

* Pregnant or breastfeeding
* Started taking birth control pills in the 6 months prior to study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to resolution of angioedema, as defined as the time interval between when the participant first noted the onset of symptoms and when there is no objective evidence of angioedema by physical examination | Measured at follow-up visit 7 days following resolution of angioedema

SECONDARY OUTCOMES:
Length of hospital stay, admission to the intensive care unit, requirement for intubation, duration of intubation, use of steroids, use of histamine receptor type 1 (H1) and H2 blockers, use of epinephrine, and blood pressure levels | Measured at follow-up visit 7 days following resolution of angioedema

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States